CLINICAL TRIAL: NCT06458751
Title: Electrophysiological Study of Berrettini Anastomosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Principal Investigator, Alberto Cappellari, Medical Doctor, Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: MANOSENS
Record Dates: First submitted 2024-05-22; First posted 2024-06-14 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Electrophysiologic Study; Hand Anastomosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 30 healthy subjects with no history of neuromuscular disease (Other): 30 healthy subjects with no history of previous neuromuscular disease and no abnormalities on neurological examination
  Interventions: Other: electrophysiological study; Device: electromyograph

INTERVENTIONS:
Other: electrophysiological study — Antidromic sensory nerve conduction studies of median and ulnar nerves will be performed on both hands of 30 healthy subjects with no history of previous neuromuscular disease and no abnormalities on neurological examination., by using surface electrical stimulation at wrist and surface digital recording electrodes on both sides of D4.
Device: electromyograph — surface electrical stimulation at wrist and surface digital recording electrodes on both sides of D4.

SUMMARY:
The common opinion that sensory supply of digit 5 (D5) and medial half of digit 4 (D4) of the hand is by ulnar nerve, while the lateral half of D4 and the remaining digits is by median nerve is an oversimplification of a complex topic. Indeed, the literature demonstrated that both the median and ulnar nerves display a number of deviations to the traditionally taught branching patterns.

The aim of our study was to investigate the physiological role of median and ulnar nerves in the sensory supply of D4.

ELIGIBILITY:
Inclusion Criteria:

* age 24-60 years
* male and female
* under informed consent
* no history of previous neuromuscular disease and no abnormalities on neurological examination

Exclusion Criteria:

-

Ages: 24 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2024-01-25 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
analysis of the sensory potential (UV amplitude in MSEC) recorded on both sides of the IV finger of the hand by stimulation of the median nerve and the ulnar one | immediately after the procedure
analysis of the sensory potential ( latency in MSEC) recorded on both sides of the IV finger of the hand by stimulation of the median nerve and the ulnar one | immediately after the procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Pediatric Emergency Department Clinica de Marchi, Foundation IRCCS Ca' Granda, Ospedale Maggiore Policlinico, Milan, Italy